CLINICAL TRIAL: NCT00186940
Title: A Study of Rasburicase Treatment for Chemotherapy of Malignancy-Induced Hyperuricemia in Patients With a History of Asthma Allergies
Brief Title: Rasburicase Treatment for Chemotherapy or Malignancy-Induced Hyperuricemia in Asthma/Allergy Patients
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: RASALL
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2011-10

CONDITIONS: Leukemia; Lymphoma; Tumor Lysis Syndrome; Hyperuricemia
Keywords: leukemia
MeSH Terms: conditions — Leukemia; Lymphoma; Tumor Lysis Syndrome; Hyperuricemia | interventions — rasburicase

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Drug: Rasburicase

INTERVENTIONS:
Drug: Rasburicase — Rasburicase 0.2 mg/kg/dose by the intravenous route for up to 7 days.

SUMMARY:
This is a multi-center trial for rasburicase in children at high risk of tumor lysis syndrome who have a history of asthma/atopy. The main purpose of this study is to establish the safety of this drug in patients with a history of asthma or severe allergies.

DETAILED DESCRIPTION:
Because they were excluded from most of the clinical trials of non-recombinant urate oxidase and rasburicase, the safety of rasburicase in this population is not known, though preliminary data indicates that the drug is safe. The primary objective of this study is to estimate the proportion of grade 3 or 4 allergic reactions to rasburicase in patients with a history of asthma or severe allergy (to antigens other than rasburicase or other urate oxidases) treated with rasburicase for the prevention or treatment of malignancy or chemotherapy-induced hyperuricemia. Patients at risk of tumor lysis syndrome with a history of asthma/atopy will be treated with rasburicase according to standard practice and observed for allergic reactions.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of hematologic malignancy.
* Existing hyperuricemia or high risk of developing hyperuricemia of malignancy.
* The treating clinician plans to treat the patient with rasburicase. A patient is only eligible for RASALL if the clinician has already decided to use rasburicase. Rasburicase should not be given in order to make a patient eligible for this non-therapeutic observational study.
* No prior exposure to rasburicase or other urate oxidase.
* A history of asthma or significant allergy.

Exclusion Criteria

* Wheezing or an active hypersensitivity reaction at entry.
* Hypersensitivity to Aspergillus proteins.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients at high risk of tumor lysis syndrome who have a history of asthma, eczema, or significant allergies (to substances other than rasburicase).
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2005-03; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Incidence of grade 3 or 4 allergic reactions | Within 30 days of last treatment administration

CONTACTS AND LOCATIONS:
Overall Officials: Raul C. Ribeiro, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (11):
- United States (11):
  - Stanford University, Palo Alto, California
  - Rady Children's Hospital, San Diego, California
  - Peyton Manning Children's Hospital at St. Vincent, Indianapolis, Indiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Children's Hospital Michigan, Detroit, Michigan
  - Columbia University Medical Center, New York, New York
  - Rhode Island Hospital, Providence, Rhode Island
  - St.Jude Children's Research Hospital, Memphis, Tennessee
  - Cook Children's Medical Center, Fort Worth, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Mid-West Children's Cancer Center, Milwaukee, Wisconsin

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org